CLINICAL TRIAL: NCT04825704
Title: Can Topical Administration of Bupivacaine Reduce Pain After Tonsillectomy?
Brief Title: Bupivacaine in Tonsillectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nordlandssykehuset HF (Other)
Responsible Party: Principal Investigator, Kristin Sandal Berg, MD PhD, Trainee in anesthesiology, associate professor, Nordlandssykehuset HF
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BupivacTons20
Record Dates: First submitted 2021-03-24; First posted 2021-04-01 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bupivacaine (Active Comparator): Topical administration of bupivacaine via gauze swab in the tonsillar fossae after removal of throat tonsils.
  Interventions: Drug: Bupivacaine
- Sodium chloride (Placebo Comparator): Topical administration of 0,9% sodium chloride via gauze swab in the tonsillar fossae after removal of throat tonsils.
  Interventions: Drug: Sodium chloride

INTERVENTIONS:
Drug: Bupivacaine — Topical administration of bupivacaine via gauze swab in the tonsillar fossae after removal of throat tonsils.
  Other Names: Marcain
  Arms: Bupivacaine
Drug: Sodium chloride — Topical administration of 0,9% sodium chloride via gauze swab in the tonsillar fossae after removal of throat tonsils.
  Other Names: Saline
  Arms: Sodium chloride

SUMMARY:
A placebo-controlled and double-blind study is planned according to current legislation and ICH GCP guidelines with 80 patients at Nordland Hospital, Bodø. Fifty percent are randomized to receive bupivacaine 5 mg / ml on the gauze swabs used to stop the bleeding after tonsillectomy, and 50% receive 0.9% sodium chloride.

Pain at rest and pain when swallowing according to numerical rating scale (0-10), as well as the presence of the following symptoms (yes / no): nausea, vomiting, food intake, bleeding, fever, need for extra painkillers in the form of morphine or similar will be registered 1, 2, 3, 4, 5, 6 hours and 1, 2 4 and 6 days after the operation. Differences are analyzed with "mixed models" statistics and the results will be published in a peer-based journal.

ELIGIBILITY:
Inclusion Criteria:

All patients undergoing isolated tonsillectomy from the age of 5 years to 40 years

Exclusion Criteria:

1. Known allergy to local anesthetics.
2. Patients using painkillers in the form of opioids fixed before inclusion in the study. People who have a lot of pain often have more pain after known painful stimuli, such as surgery. This is known as the phenomenon of "central sensitization" and "opioid-induced hyperalgesia" and will probably contribute to great heterogeneity within the groups. Because very few people use opioids regularly from those who have an isolated tonsillectomy performed, it can make it difficult to detect any differences between the groups, and the number is far too low to be able to perform stratified analyzes on only these people.
3. Persons weighing less than 10 kg.
4. Persons over the age of 18 who are not competent to give consent.
5. Patients using class Ib antiarrhythmics (lidocaine, mexiletine) due to increased risk of additive toxicity due to structural similarities. (see SPC)
6. Known partial or total heart block that has not had a pacemaker inserted (see SPC)
7. Severe hepatic failure (spontaneous prothrombin time -international normalized ratio (PT-INR)> 2.0). These patients are not offered this type of procedure as day surgery due to the high risk of complications for the surgery itself.
8. Severe renal failure (estimated glomerular filtration rate <15 ml / min / 1.73m2).

Ages: 5 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 84 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2023-06-27 (Actual)

PRIMARY OUTCOMES:
Difference in self-reported pain at rest. | Until 6 hours postoperatively.
  Difference in self-reported pain at rest by the numerical rating scale (0-10, 0 = no pain, 10 worst pain) for patients aged 10 years and older, and indicated by the faces pain scale-revised (0-10, 0 = no pain, 10 worst pain) for patients aged 5-10 years old, on average over all measurement times. Pain is registered at 1,2,3,4,5 and 6 hours.

SECONDARY OUTCOMES:
Difference in pain when swallowing on average over all measurement times. | Until 6 days postoperatively
  Difference in pain according to the numerical rating scale (0-10, 0 = no pain, 10 worst pain) between the two groups when swallowing on average over all measurement times. Pain is registered at 1,2,3,4,5 and 6 hours, and 1,2,4 and 6 days postoperatively.
Graphic Descriptive representation of numerical rating scale (0-10, 0 = no pain, 10 worst pain) in a curve diagram | Until 6 days postoperatively
  Pain is registered at 1,2,3,4,5 and 6 hours, and 1,2,4 and 6 days postoperatively
Difference in numerical rating scale (0-10, 0 = no pain, 10 worst pain) at rest between the groups day 1 after the operation | Until 1 day postoperatively
Difference in numerical rating scale (0-10, 0 = no pain, 10 worst pain) at rest between the groups day 6 after the operation | Until 6 days postoperatively
Difference in numerical rating scale (0-10, 0 = no pain, 10 worst pain) when swallowing between the groups day 1 after the operation | Until 1 day postoperatively
Difference in numerical rating scale (0-10, 0 = no pain, 10 worst pain) when swallowing between the groups day 6 after the operation | Until 6 days postoperatively
Difference in defined daily doses of morphine in the two groups | Until 6 days postoperatively
Difference in number and type a) serious adverse event, b) serious adverse reaction and c) adverse reaction where the adverse reaction is an adverse medical event where there is a probable or possible association with the test preparation | Until one hour postoperatively
Difference in hours of nausea | Until 6 days postoperatively
Difference in the number of times eaten solid food | Until 6 days postoperatively
Number of vomiting episodes | Until 6 days postoperatively
Number of episodes in which blood is spit for more than 30 minutes from 1 hour postoperatively | Until 6 days postoperatively
Hours with measured fever> = 38 C rectally, tympanometric or with temporal scanner | Until 6 days postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Kristin S Berg, MD PhD, Principal Investigator — Nordlandssykehuset HF; Erik W Nielsen, MD PhD, Principal Investigator — Nordlandssykehuset HF
Locations (1):
- Nordland Hospital, Bodø, Norway